CLINICAL TRIAL: NCT01512004
Title: Phase III Study of Propiverine Hydrochloride Extended-Release Capsule in the Treatment of Overactive Bladder (OAB) in Chinese Population With Urgent Micturition, Frequent Micturition and/or Urge Urinary Incontinence
Brief Title: Propiverine Hydrochloride Extended-Release Capsule for Overactive Bladder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Collaborators: APOGEPHA Arzneimittel GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LEES-MIC
Record Dates: First submitted 2010-11-24; First posted 2012-01-19 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Overactive Bladder
Keywords: Overactive Bladder; urgent micturition; frequent micturition; urge urinary incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge | interventions — propiverine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propiverine Hydrochloride Extended-Release Capsule (Active Comparator): 30 mg/capsule; oral; once per day
  Interventions: Drug: Propiverine Hydrochloride
- Tolterodine Extended-release Tablet (Placebo Comparator): 4mg/tablet; oral; once per day
  Interventions: Drug: Tolterodine Extended-release Tablet

INTERVENTIONS:
Drug: Propiverine Hydrochloride — drug of oral capsule
  Other Names: Mictonorm; Propierine Hydrochloride Extended-Release Capsule
  Arms: Propiverine Hydrochloride Extended-Release Capsule
Drug: Tolterodine Extended-release Tablet — 4mg/tablet; oral; once per day
  Arms: Tolterodine Extended-release Tablet

SUMMARY:
The purpose of this Phase III study is to evaluate the efficacy and safety of Propiverine Hydrochloride Extended-Release Capsule in the treatment of overactive bladder in Chinese population with urgent micturition, frequent micturition and/or urge urinary incontinence.

DETAILED DESCRIPTION:
This is a multi-center, randomized, doubled-blind, double dummy clinical study, in comparison with Tolterodine Tartrate Extended-Release Tablet as active parallel control to evaluate the efficacy and safety of Propiverine Hydrochloride Extended-Release Capsule in the treatment of Overactive Bladder in Chinese population with urgent micturition, frequent micturition and/or urge urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65, male or female patient has a diagnosis of overactive bladder and the symptoms of OAB>3 months subject has urinary frequency (average micturition frequency within 24h>8 times), urgency and/or urge incontinence by micturition diary card during screening period
* Mean volume of single micturition is less than 200ml by micturition diary dard during screening period
* The subject is willing and able to complete the micturition diary card correctly
* Subject's urine routine test show that he/she has no urinary tract infection Subject signs informed consent form

Exclusion Criteria:

* Confirmed by the investigator that subject has severe stress incontinence.
* Subject who has serious heart disease or arrhythmia, in the investigator's opinion, is not suitable to enroll.
* Subject who has contraindications of anticholinergic therapy, such as urinary retention, gastric retention and uncontrollable angle closure glaucoma.
* Subject who has a symptomatic acute urinary tract infection.
* Subject who has a recurrent urinary tract infection.
* Subject who has interstitial cystitis.
* Subject who has an agnogenic hematuria.
* Subject who has a bladder outlet obstruction of clinical significance.
* Subject who needs retention catheterization or intermittent catheterization.
* Patient with malignant tumor.
* Subject who has received anticholinergic drugs or other drugs for treating OAB within washout period, or who will receive these drugs after this study begins.
* Subject who is pregnant or lactating, or plans to be pregnant subject who has received other clinical study drugs or its participating in other clinical trial within 30 days.
* Women of childbearing age who has not taken sufficient contraception measures within 3 months before random number distribution; or intends to stop the contraception measures during the trial or within one month after the treatment is over.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2010-01; Primary Completion 2010-01 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Alteration of mean micturition frequency within 24h on the basis of continuous 3-day record | prior to medication and 8 weeks after medication
  The voiding frequency per 24 hours, and the alteration of mean micturition frequency within 24 hours on the basis of continuous 3-day record, prior to medication and 8 weeks after medication

SECONDARY OUTCOMES:
The alteration of mean incontinence frequency and mean micturition frequency and volume within 24 hours on the basis of continuous 3-day record | prior to medication, 2 weeks and 8 weeks after medication
  The alteration of mean incontinence frequency, mean micturition frequency and volume within 24 hous on the basis of continuous 3-day record,prior to medication, 2 weeks and 8 weeks after medication. Additionaly, to evaluate the subject's feeling of treatment benefit and the time of the drug effect onset.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Li, PhD, Study Director — Lee's Pharmaceutical
Locations (1):
- Beijing Chaoyang Hospital, Beijing, China